CLINICAL TRIAL: NCT04942717
Title: Communicating With Oncology Nurses About Values From the Outset (CONVO): An Innovative Primary Palliative Care Intervention in English and Espanol
Brief Title: Adapting for Latinx Populations an Intervention That Involves Discussing and Sharing Patients' Health-Related Values
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 20-539
Record Dates: First submitted 2021-06-21; First posted 2021-06-28 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Solid Tumor; Solid Tumor, Adult; Solid Tumor, Unspecified, Adult
Keywords: Spanish speaking; Latinx; Solid Tumor; 20-539; Memorial Sloan Kettering Cancer Center

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aim 1 (Experimental): For the survey component, recruitment will focus on patients who have not participated in a semi-structured interview as part of the Aim 1 research. For Aim 1, we will seek to recruit approximately 36 patients and 12 family members for the initial key informant interviews, 20 patients for the followup survey, and 10 for the English/backtranslated-English side-by-side comparison.
  Interventions: Behavioral: CONVO intervention
- Aim 2 (No Intervention): Patients who provide consent during Months 9-11 (i.e., first three months of "Control Period" of pilot trial) will be in the "control group," with follow-up for outcomes data collection occurring during Months 12-14. Patients who provide consent during Months 16-18 (after implementation of the intervention at the end of Month 15) will be in the "intervention group" and will be followed for three more months (Months 19-21) for outcomes data collection. We will enroll a total of 130 patients (65 in control period, 65 in intervention period) during the pilot trial across the two trial sites, SBH and Jacobi, to reflect, as much as possible, the relative patient numbers and the demographic composition of the sites. During the intervention period, family who accompany patients to clinic and are included (patient option to include one family member) in the CONVO values discussions will be approached (in person or via video conferencing platform or telephone) for participation at the clinic.

INTERVENTIONS:
Behavioral: CONVO intervention — The CONVO intervention consists of oncology nurse-led discussions exploring patients' health-related values as part of routine oncology care for all patients, from the beginning of oncologic care. Nurses will use the Nurse's Values Discussion Guide. At these sites, chemotherapy nurses will deliver the CONVO discussion, as patients at these sites do not have primary nurses assigned and because oncology doctors, BPs and PAs do not work one-on-one as a pair with a unique nurse.
  Arms: Aim 1

SUMMARY:
The purpose of this study is to translate and tailor for Latinx participants a program called Communicating with Oncology Nurses about Values from the Outset (CONVO). In CONVO, routine cancer care for each participant includes a discussion between the nurse and participant about the participant's health-related values.

ELIGIBILITY:
Inclusion Criteria:

* All participants will be adults (age ≥ 21) providing informed verbal consent. We seek a waiver of signed consent, which will allow use of virtual communication during the COVID-19 pandemic period.
* Patients will be eligible as key informants in the translation/transcreation process (Aim 1) if they are receiving medical oncology care for a solid tumor malignancy at RLC, SBH, or Jacobi and speak Spanish as their preferred language. In addition, English-speaking Latinx patients will be eligible to participate in interviews based on the back-translated (Spanish-to-English) version of the Guide

  * We are focusing on patients with solid tumors rather than hematologic malignancies because 1) patients in the latter group may be receiving initial oncologic treatment in the hospital, whereas our study staff will be based at a distance from the hospital in the ambulatory clinics; 2) the trajectory, patient characteristics, and other aspects of hematologic malignancies tend to be different from solid tumor malignancies such that it would be more difficult to understand the overall impact of the intervention if patients with both types of malignancies w ere included.
* Spanish-speaking family/other informal caregivers (collectively referred to as "family") who accompany participating patients to clinic will also be eligible to participate in interviews as part of the Aim 1 translation/transcreation process. These will be individual interviews, conducted separately for patient and family participants.
* Clinicians eligible for participation in the transcreation will be oncology physicians, nurses and other key clinical staff (e.g. social workers, advance practice providers, etc.) at RLC and other MSK sites who are Latinx and/or whose practice includes >20% Latinx patients.
* Site leaders at SBH, Jacobi, and RLC with administrative responsibility for medical oncology will be eligible as key informants in transcreation of CONVO.
* For the Aim 2 pilot trial, patients will be eligible if they are receiving systemic chemotherapy at SBH or Jacobi for a solid tumor; identify as Latinx; and speak English and/or Spanish. Family and/or informal caregivers who accompany the patient and speak English and/or Spanish will also be eligible (if the patient opts to include the family and/or informal caregiver in the CONVO discussion).
* Nurses providing outpatient oncology care in chemotherapy areas at SBH or Jacobi will be eligible to participate in the pilot trial.

Exclusion Criteria:

* Inability to understand consent procedure in either English or Spanish will be an exclusion. (The consenting professional will be bilingual [English/Spanish] and able to explain and obtain consent in either language.)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Estimated)
Dates: Start 2021-06-18 (Actual); Primary Completion 2026-06-18 (Estimated); Study Completion 2026-06-18 (Estimated)

PRIMARY OUTCOMES:
Translation/transcreation of the CONVO intervention | 24 months
  To translate/transcreate (linguistic plus cultural adaptation) our intervention for implementation with Spanish-speaking Latinx cancer patients receiving outpatient oncologic care in their communities: Comunicar Nuestros Valores a las enfermeras de Oncología desde el comienzo del tratamiento de cáncer.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Nelson, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (5):
- United States (5):
  - MSK at Ralph Lauren (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - SBH Health System, The Bronx, New York
  - Jacobi Medical Center, The Bronx, New York
  - New York Cancer & Blood Specialists (Data collection only), The Bronx, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org